CLINICAL TRIAL: NCT02988882
Title: A Multi-Center, Randomized, Double-Masked, Vehicle Controlled Phase 3 Study Evaluating the Efficacy and Safety of OTX-DP for the Treatment of Chronic Allergic Conjunctivitis Using a Modified Conjunctival Allergen Challenge Model (CAC®)
Brief Title: OTX-15-002: A Phase 3 Study Evaluating the Safety and Efficacy of OTX-DP for the Treatment of Chronic Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-15-002
Record Dates: First submitted 2016-12-02; First posted 2016-12-09 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2018-03

CONDITIONS: Chronic Allergic Conjunctivitis
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- OTX-DP (Experimental): OTX-DP (dexamethasone insert) 0.4 mg for intracanalicular use
  Interventions: Drug: Dexamethasone
- PV (Placebo Comparator): PV (placebo drug delivery vehicle)
  Interventions: Other: Placebo Vehicle

INTERVENTIONS:
Drug: Dexamethasone
  Arms: OTX-DP
Other: Placebo Vehicle
  Arms: PV

SUMMARY:
The objective of the study was to evaluate the efficacy and safety of OTX-DP (dexamethasone insert) 0.4 mg for intracanalicular use when placed in the canaliculus of the eyelid for the treatment of the signs and symptoms of chronic allergic conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Has a positive history of ocular allergies and a positive skin test reaction to a perennial allergen and a seasonal allergen
* Has a positive bilateral CAC reaction to a perennial allergen within minutes of instillation

Exclusion Criteria:

* History of refractive surgery (including LASIK procedures) within the past 2 years
* History of retinal detachment, diabetic retinopathy, or active retinal disease
* Presence of an active ocular infection or positive history of an ocular herpetic infection at any visit
* Use any of the disallowed medications during the period indicated
* History of IOP increase as a result of steroid treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04-27 (Actual); Study Completion 2016-04-27 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Vehicle: PV (placebo drug delivery vehicle)
Period: Overall Study
Arm/Group | OTX-DP | Placebo Vehicle
Started | 44 | 42
Completed | 41 | 40
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OTX-DP | Placebo Vehicle | Total
Number analyzed (Participants) | 44 | 42 | 86
Age, Continuous [Mean (Full Range); unit: years] | 39.1 [20 to 68] | 42.2 [18 to 70] | 40 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 18 | 17 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 21
  Not Hispanic or Latino | 33 | 32 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 35 | 40 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Iris Color [Count of Participants; unit: Participants]
  Black | 1 | 0 | 1
  Blue | 6 | 15 | 21
  Brown | 24 | 19 | 43
  Hazel | 5 | 3 | 8
  Green | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching Post-CAC (Conjunctival Allergen Challenge) at Visit 6
Description: Modified CAC model (Ora, Andover, MA); Grade 0-4, allowing half unit increments; 0=No itching
Time Frame: 3 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 44 | 42
units on a scale | 2.04 (1.088) | 2.31 (1.115)

2. Primary Outcome: Ocular Itching Post-CAC (Conjunctival Allergan Challenge) at Visit 6
Description: Modified CAC model (Ora, Andover, MA); Grade 0-4, allowing half unit increments; 0=No itching
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 44 | 42
units on a scale | 2.07 (1.100) | 2.41 (1.039)

3. Primary Outcome: Ocular Itching Post-CAC (Conjunctival Allergen Challenge) at Visit 6
Description: Modified CAC model (Ora, Andover, MA); Grade 0-4, allowing half unit increments; 0=No itching
Time Frame: 7 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTX-DP | Placebo Vehicle
Number analyzed (Participants) | 44 | 42
units on a scale | 2.02 (1.131) | 2.37 (1.129)

ADVERSE EVENTS:
Arm/Group | OTX-DP | Placebo Vehicle
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 6/41 | 11/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTX-DP (N=41) | Placebo Vehicle (N=40)
Adverse Events (General disorders) | 6 (7) | 11 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No